CLINICAL TRIAL: NCT03545230
Title: Four "Not" Technique in Delayed and Nonunion of Lateral Humeral Condyle Fracture in
Brief Title: Results of "Four Not Techniques" in Delayed and Nonunion Fractures of Lateral Humeral Condyle in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si 355/2016
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Orthopaedic Surgery

STUDY DESIGN:
Intervention Model Description: all childre with delayed union and nonunion lateral humeral condyle will be included.
  After informed consent and full explanation.The Four Not Techniques""will be done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children who recieved "Four Not Techniques" surgery (Experimental): :Four Not Techniques"
  Interventions: Procedure: :Four Not Techniques"

INTERVENTIONS:
Procedure: :Four Not Techniques" — :Four Not Techniques"
  1. Not enter posteriorly
  2. Not too much dissection the muscle around the lateral condyle during surgery
  3. Not perfect anatomical reduction
  4. Not using bone graft.

SUMMARY:
Fracture of lateral humeral condyle in children is not uncommon.The nonunion means no healing of the fracture after 3 months from the injury.Delayed union means no healing from 6 weels to less than 3 months after injury.

The treatment is difficult even surgery because of lack of blood supply of lateral condyle,unstability from muscle force and the articular fluid inhibition of union.

The author try to improve the healing of the fracture after surgery by "4 not techniques",

1. the surgical approach should not enter posteriorly because the blood supply of lateral condyle enter posteriorly in order to avoid cut the vessels.
2. The dissection should not too much especially the muscle around the condyle.
3. It is not necessary to perfectly reduced the fracture after nonunion to avoid too much dissection the muscle and allow only healing of the fragment.
4. Bone graft is not necessary. The author wants to know the results after perform "4 not technique" in delayed union and nonunion of lateral humeral condyle fracture

DETAILED DESCRIPTION:
All children with delayed union or nonunion fracture lateral humeral condyle fractures will be inclued in the study.

The children who received the previous surgery of the same elbow will be excluded.

After full explanation and discussion to the children and parents.The surgery in "4 not technique" will be performed.

1. the lateral approach of the affected elbow and enter the fracture anteriorly. The approach should not enter posteriorly because the blood supply of lateral condyle enter posteriorly in order to avoid cut the vessels.
2. The dissection should not too much especially the muscle around the condyle. The nonunon fragment will be cleaned,washed and made until the healthy bone surface of fracture appear in both side of fracture.
3. It is not necessary to perfectly reduced the fracture after nonunion to avoid too much dissection the muscle and allow only healing of the fragment.The fixation by K-wires or screw in older children until the fragment is stable enough.
4. Bone graft is not necessary but in valgus deformity the correctuve osteotomy should be performed to correct the valgus.

The skin is closed,the long arm cast is put and change in 2 weeks interval until bone union.

The measurement will be

1. The union rate
2. The carrying angle , Baumann angle,shaft condylar angle
3. ROM
4. Complication of surgery such as infection,AVN of troclear etc.

ELIGIBILITY:
Inclusion Criteria:

* all children less than 18 years old with delayed union and nonunion of fracture lateral humeral condyle

Exclusion Criteria:

* any previous surgery at the same elbow
* refuse to participate the research

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06-10 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
the union rate | 1 year
  the healing of the fracture in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Kamolporn Kaewpornsawan, MD., Principal Investigator — Department of Orthopaedic Surgery,Faculty of Medicine,Siriraj Hospital,Mahidol University,Bangkok,Thailand
Locations (1):
- Faculty of Medicine Siriraj Hospital Mahidol University, Bangkok, Thailand